CLINICAL TRIAL: NCT01583270
Title: Effect of Arabinoxylan and Rye Kernels on Second Meal Responses in Subjects With the Metabolic Syndrome
Brief Title: Effect of Arabinoxylan and Rye Kernels on Second Meal Responses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Collaborators: University of Aarhus (Other)
Responsible Party: Principal Investigator, AnneMarie Kruse, Professor Kjeld Hermansen, Aarhus University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: CERN-biofuncarb second meal; 2101-08-0068 (Other Grant/Funding Number: Danish council for strategic research)
Record Dates: First submitted 2012-04-18; First posted 2012-04-24 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Metabolic Syndrome
Keywords: Arabinxylan; Rye kernels; whole grain; Dietary fibre; Metabolic syndrome; Glycemic response; Colon fermentation; Second meal effekt; Satiety
MeSH Terms: conditions — Metabolic Syndrome | interventions — arabinoxylan; Dietary Fiber; Flour

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arabinoxylan (Experimental): Porridge rich in arabinoxylan. 50 g available carbohydrate
  Interventions: Dietary Supplement: Arabinoxylan
- rye kernels (Experimental): Porridge made from rye kernels. 50 g available carbohydrate
  Interventions: Dietary Supplement: Rye kernel
- arabinoxylan and rye kernels (Experimental): Porridge made of rye kernels and arabinoxylan. 50g available carbohydrate
  Interventions: Dietary Supplement: Arabinoxylan and rye kernels
- semolina (Experimental): Semoline porridge. 50 g available carbohydrate
  Interventions: Dietary Supplement: Semolina

INTERVENTIONS:
Dietary Supplement: Arabinoxylan — Porridge rich in arabinoxylan
  Other Names: Dietary fibre.
  Arms: Arabinoxylan
Dietary Supplement: Rye kernel — Porridge made of rye kernels
  Other Names: Whole grain. Rye. Kernels.
  Arms: rye kernels
Dietary Supplement: Arabinoxylan and rye kernels — Porridgde made of rye kernels and arabinoxylan
  Other Names: dietary fibre. whole grain. rye kernels.
  Arms: arabinoxylan and rye kernels
Dietary Supplement: Semolina — Semoline porridge. control meal.
  Other Names: Wheat.
  Arms: semolina

SUMMARY:
Sedentary lifestyles and increasing obesity are main causes of the global increase in the prevalence of the metabolic syndrome (Mets) and type 2 diabetic (T2DM). Diet quality, particularly composition of carbohydrate play also a significant role. Barley, oat and rye may in addition to reducing the acute post prandial glucose response also reduce glucose response at a subsequent meal. Purified dietary fibre has been shown to reduce GI and affect levels of satiety hormones. In contrast, our knowledge of the physiological effect of arabinoxylan, which constitute a substantial part of dietary fibre in cereal products, is limited in relation to second meal effects. The investigators also lack knowledge of the second meal effect of arabinoxyan in combination with rye kernels.

Hypothesis: Porridge rich in arabinoxylan and/or whole rye kernels can increase the formation of short chain fatty acids and improve the glycemic response.

The aim of the present study is to compare the effect of porridge test meals based on purified arabinoxylan, rye kernels, a combination of arabinoxylan and rye kernels, and semolina porridge as control on acute postprandial response as well as response at a subsequent standardized meal. The study will be conducted in subjects with the metabolic syndrome. The primary endpoint is glucose response. Secondary endpoints are the following items: insulin, incretins, inflammatory markers, ghrelin, free fatty acids, metabolomics, breath hydrogen and subjective satiety feeling.

This project will improve opportunities for identifying and designing foods with low GI that is particularly suited to people who are at high risk of developing T2DM. The investigators also expect to gain a greater understanding of the metabolic fingerprint, as seen after ingestion of low-GI foods and thereby gain a molecular understanding of how low-GI foods affect health by altering metabolic processes. This will give us a deeper insight into the metabolic processes that are necessary for maintaining normal glucose homeostasis

DETAILED DESCRIPTION:
Using a cross-over design, 15 subjects with Mets will consume test meals containing four different porridges in randomized order. Blood samples will be collected over 2 hours after ingestion of test meals and 2 hours after ingestion of a standard second lunch meal served 4 hours after the test meals. The amount of porridge and the standard lunch are equivalent to 50 g available carbohydrate. Visual Analog Scale (VAS) will be used for determination of subjective satiety feeling and measurements of breath hydrogen will be used as a marker for colon fermentation.

ELIGIBILITY:
Inclusion Criteria:

Central obesity (Female > 94 cm; Male > 80 cm) with two of the following:

1. fasting triglyceride (> 1,7 mmol/L),
2. HDL-cholesterol: (Female:< 1,03 mmol/L; Male:< 1,29 mmol/L),
3. blood pressure (≥ 130/85 mmHg) and
4. fasting plasma glucose (≥ 5,6 mmol/L)). Subjects who are in medical treatment with lipid and blood pressure-lowering drugs can continue with their habitual treatment provided that the treatment is stable throughout the trial.

Exclusion Criteria:

* fasting plasma glucose > 7,0 mmol/l,
* fasting plasma triglyceride > 5,0 mmol/l,
* blood pressure > 160/100 mmHg ,
* legal incapacity , endocrine, cardiovascular or kidney disease,
* BMI > 38kg/m2,
* corticosteroid treatment,
* alcohol or drug addiction and
* pregnancy or lactation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2012-04; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Glucose response after second meal | 2 hours

SECONDARY OUTCOMES:
Plasma response after second meal | 2 hours
  Plasma insulin, incretins, ghrelin, short chain fatty acids, freee fatty acids, inflammation markers, and metabolomics.
Plasma response after test meal | 2 hours
  Plasma glucose, insulin, incretins, short chain fatty acids, free fatty acids, metabolomisc.
Breath hydrogen after second meal | 2 hours
  Breath hydrogen as marker for colon fermentation
Breath hydrogen after testmeal | 2 hours
  Breath hydrogen as marker for colen fermentation
Satiety feeling after second meal | 2 hours
Satiety feeling after test meal | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Kjeld Hermansen, Professor, Principal Investigator — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Aarhus, Denmark